CLINICAL TRIAL: NCT04045301
Title: A 15 Months, Double-Blind, Randomized Controlled Trial Comparing 20 Weeks of Two Dosages of Omalizumab to Placebo to Accelerate a Symptom-driven Oral Immunotherapy Schedule in Subjects Aged 6 to 25 Years With Multiple Food Allergies
Brief Title: Omalizumab to Accelerate a Symptom-driven Multi-food OIT
Acronym: BOOM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Philippe Bégin (Other)
Collaborators: The Hospital for Sick Children (Other); Centre hospitalier de l'Université de Montréal (CHUM) (Other); Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Sponsor-Investigator, Philippe Bégin, Principal Investigator, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITO-OMA-2018-01
Record Dates: First submitted 2018-11-30; First posted 2019-08-05 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Food IgE-mediated Allergy; Immunotherapy; Omalizumab; Physiological Effects of Drugs
Keywords: multi-food OIT; oral immunotherapy; omalizumab; symptom-driven protocol; double-Blind, randomized controlled trial
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Omalizumab 16 mg/kg (Experimental): Participants will receive omalizumab 16 mg/kg monthly doses for 12 weeks, followed by omalizumab 8 mg/kg monthly for 4 weeks and then omalizumab 4 mg/kg monthly for 4 weeks.
  Multi-food oral immunotherapy following a symptom-driven schedule will begin 8 weeks after starting study drug.
  Interventions: Biological: Omalizumab 16mg/kg; Other: Multi-food oral immunotherapy (OIT)
- Omalizumab 8 mg/kg (Experimental): Participants will receive omalizumab 8 mg/kg monthly doses for 12 weeks, followed by omalizumab 4 mg/kg monthly for 4 weeks and then omalizumab 2 mg/kg monthly for 4 weeks.
  Multi-food oral immunotherapy following a symptom-driven schedule will begin 8 weeks after starting study drug.
  Interventions: Biological: Omalizumab 8mg/kg; Other: Multi-food oral immunotherapy (OIT)
- Placebo (Placebo Comparator): Participants will receive placebo doses for 20 weeks. The doses will be injected every 2 or 4 weeks depending on the weight of the participant.
  Multi-food oral immunotherapy following a symptom-driven schedule will begin 8 weeks after starting study drug.
  Interventions: Biological: Placebo; Other: Multi-food oral immunotherapy (OIT)

INTERVENTIONS:
Biological: Omalizumab 16mg/kg — Participants will receive omalizumab 16 mg/kg monthly doses for 12 weeks, followed by omalizumab 8 mg/kg monthly for 4 weeks and then omalizumab 4 mg/kg monthly for 4 weeks, for a total of 20 weeks including a taper period.
  Arms: Omalizumab 16 mg/kg
Biological: Omalizumab 8mg/kg — Participants will receive omalizumab 8 mg/kg monthly doses for 12 weeks, followed by omalizumab 4 mg/kg monthly for 4 weeks and then omalizumab 2 mg/kg monthly for 4 weeks, for a total of 20 weeks including a taper period.
  Arms: Omalizumab 8 mg/kg
Biological: Placebo — Participants will receive placebo for 8 weeks prior to the initiation of oral immunotherapy and 12 weeks after for a total of 20 weeks including a taper period.
  Arms: Placebo
Other: Multi-food oral immunotherapy (OIT) — Multi-food oral immunotherapy will be conducted to a mix of three foods. It will be started 8 weeks after study drug with an initial food escalation. Participants will undergo biweekly increase until they tolerate a maintenance dose of 1500 mg (500 mg per food) of food protein.

SUMMARY:
This study will determine the dose-related efficacy of a 20-week treatment of omalizumab started 8 weeks before the onset of a symptom-driven multi-food oral immunotherapy (OIT) protocol at decreasing time to OIT maintenance dose. Two dosages of omalizumab will be compared to placebo during an oral immunotherapy protocol for three simultaneous food allergens.

DETAILED DESCRIPTION:
This is a phase 2b, multi-center randomized controlled trial comparing 2 doses of omalizumab to placebo in subjects 6 to 25 years old with multiple food allergies undergoing a symptom-driven multi-food OIT protocol.

Subjects will undergo a screening period involving a DBPCFC to a mix of three allergens which will determine their eligibility and eliciting dose.

Eligible subjects will be randomized to one of 2 omalizumab dosages or placebo at a ratio of 2:2:1 for a total period of 20 weeks.

They will undergo initial food escalation (IFE) to determine their starting food treatment mix dose for three simultaneous food allergens after a pre-treatment period of 8 weeks with the study drug.

Subjects will undergo up-dosing OIT visits at the clinic every two weeks, until a maintenance dose of 1500mg of protein (500mg per food) is reached (primary endpoint).

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects 6 to 25 years old at screening visit.
2. History of IgE-mediated allergy to at least three foods within the following list: peanut, milk, egg, wheat, oat, soy, barley, rye, buckwheat, hazelnut, pecan, cashew, pistachio, almond, walnut and sesame.
3. Subjects currently following a strict avoidance of these three foods.
4. Positive SPT with a largest wheal diameter ≥ 6 mm to all three foods.
5. Food-specific IgE level greater than 15 kU/L for all three foods
6. Positive DBPCFC to treatment food mix with an eliciting dose ≤ 300 mg of total food protein.
7. Signed informed consent and assent.

Exclusion criteria

1. Subjects reacting objectively to the placebo during the screening DBPCFC.
2. Severe asthma as defined by GINA 201948.
3. Active or past confirmed eosinophilic oesophagitis.
4. Subject currently under allergen immunotherapy.
5. Subject/parent with excessive anxiety unlikely to cope with study conditions as per investigator's opinion.
6. Subject/parent unwillingness to comply with study requirements.
7. Subject unwillingness to ingest a daily food dose of up to 1500 mg of allergen protein.
8. Inability to discontinue anti-histamine medication prior to study procedures.
9. Known allergy to omalizumab or its excipients.
10. Known allergy to components of the placebo food treatment mix that cannot be substituted without interfering with the blind (e.g.: dates, banana, chocolate syrup)
11. Use of immunosuppression or immunomodulatory drug (including omalizumab) or food oral immunotherapy or investigational treatment or procedure within 1 year.
12. Relative contraindication or inability to use epinephrine auto-injector.
13. Subjects receiving beta-blockers or angiotensin converting-enzyme (ACE) inhibitors.
14. Pregnancy or lactation for the duration of the study.
15. Any condition that is not compatible with the study treatment or procedures as per investigator judgment.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of omalizumab at decreasing time-to-maintenance during a symptom-driven multi-food OIT protocol. | Assessed up to 52 weeks after IFE
  Time from IFE to target multi-food protein maintenance dose of 1500 mg of total food protein

SECONDARY OUTCOMES:
Change in reactivity threshold to food treatment mix after pre-treatment with study drug. | Measured 8 weeks after starting investigational product
  Measured as the amount of food allergen eliciting an objective allergic reaction on double-blinded oral food challenge or initial food escalation.
Average up-dosing speed while on study drug. | From week 0 to week 12 post IFE
  Average of (log of escalation %)/(days since last escalation) for all escalation visits while on study drug
Mean cumulative function of allergic adverse events attributable to food dosing throughout the trial. | For one year following IFE
  AEs will be captured using the daily dosing diary throughout the trial, including during maintenance. Any systemic reaction having occurred since the last visit will be reviewed and graded by the investigator according to the CoFAR grading system.
Rate of treatment failure | At any time during the 12-month OIT phase
  Subject which stop daily ingestion of food treatment mix, prior to achieving study maintenance dose, for a period of 14 days or more

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bégin, MD, PhD, Principal Investigator — St. Justine's Hospital
Locations (3):
- Canada (3):
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - CIUSSS de l'Estrie - Centre Hospitalier Universitaire de Sherbrooke (CHUS), Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Langlois A, Lavergne MH, Leroux H, Killer K, Azzano P, Paradis L, Samaan K, Lacombe-Barrios J, Masse B, Des Roches A, Begin P. Protocol for a double-blind, randomized controlled trial on the dose-related efficacy of omalizumab in multi-food oral immunotherapy. Allergy Asthma Clin Immunol. 2020 Apr 17;16:25. doi: 10.1186/s13223-020-00419-z. eCollection 2020. PMID 32328115